CLINICAL TRIAL: NCT05008380
Title: Open-label, Controlled, Randomized Clinical Trial on the Efficacy of Early Prone-positioning in Patients With Mild Pneumonia Due to SARS-CoV-2
Brief Title: Efficacy of the Early Prone-positioning in Hospitalized Patients With Mild Covid-19 Pneumonia
Acronym: EpCOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Paolo Bonfanti, Director of Infectious Diseases Department, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3772
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care + prone positioning (Experimental): Standard of care. Prone-positioning cycles as the following: 3-6 hours of prone-positioning twice a day.
  Interventions: Procedure: prone positioning
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Procedure: prone positioning — 3-6 hours of prone-positioning twice a day
  Arms: Standard of care + prone positioning

SUMMARY:
The study aims to evaluate if the early prone-positioning in awake patients with mild Covid-19 pneumonia can reduce the need of high-flow oxygen-therapy, invasive or non-invasive ventilation and prevent the worsening of clinical conditions.

Patients will be randomized on a 1:1 ratio and stratified based on the onset of symptoms (<10 days; >10 days) and need of oxygen therapy (no need; need).

One branch of patients (interventional) will undergo standard of care treatment + prone-positioning cycles, the other one (controll) will undergo standard of care treatment alone.

Patients will be evaluated evaluated on the day of the enrolment, on day 1, day 3, day 7 and every 7 days until the patient dismissal or until day 28 (whichever occurs first).

Adverse events and concurrent medications will be noted as well.

The analysis will be conducted according to "intention to treat" criteria; primary outcomes will be calculated using survival-based methods.

DETAILED DESCRIPTION:
In this prospective, unicentred, open, controlled study, patients will be randomized on a 1:1 ratio using casual permutation blocks, identifying two branches of treatment: standard of care; standard of care + prone positioning. Patients will be stratified in 4 strata based on the onset of symptoms (<10 days; >10 days) and need of oxygen therapy (no need; need).

In order to obtain statistical significance, the sample size will include 96 patients.

Patients in the SOC + prone-positioning branch will undergo cycles of prone-positioning following this scheme: 3-6 hours of prone-positioning twice a day. The actual length of the cycles will be registered during the study.

Data will be collected using a dedicated CRF, which will include recording of adverse events and concurrent medications.

Patients will be evaluated on the day of the enrolment, on day 1, day 3, day 7 and every 7 days until the patient dismissal or until day 28 (whichever occurs first). If dismissal occurs before day 28, a follow-up interview will be conducted in presence or on the phone to collect the remaining data.

The analysis will be conducted according to "intention to treat" criteria; primary outcomes will be calculated using survival-based methods (Kaplan-Meier curves with log-rank test and Cox regression), while secondary outcomes will be evaluated using both survival-based methods and proportional odds model.

The occurrence of adverse events and the causes of withdrawal from the study in the two branches of treatment will be compared using chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* positive PCR for Sars-Cov-2 Rna on any respiratory samples within 7 days from enrollment
* imaging positive for pulmonary involvement or clinical evidence of respiratory involvement ( new onest of hypoxemia with 02 <80mmHg or SpO2 < 94% in air or need for oxygen therapy in oreder to mantaine SpO2 > 93%.
* need of hospitalization

Exclusion Criteria:

* start of prone-positioning cycles before being enrolled in the study
* SpO2/FiO2 <200
* need of high-flow oxygen therapy (HFNC) or need of non-invasive ventilation and/or CPAP or indications for intubation and mechanical ventilation
* relative or absolute contraindications for prone positioning (eg facial fractures, advanced pregnancy, mental status alterations, spinal instability...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Accomplishment of the end-points | 0-28 days
  the occurence of the first of the following end-points: death, start of high flow oxygen therapy, CPAP, meccanichal ventilation, P/F <200

SECONDARY OUTCOMES:
time of recovery | 0-28 days
time of weaning from oxygen | 0-28 days
variation of the clinical condition | 0-28 days
mortality | 0-28 days
number of adverse event | 0-28 days
number and duration of prone positioning cycles | 0-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonfanti, Principal Investigator — asst-monza Ospedale San Gerardo
Locations (1):
- Asst-Monza Ospedale San Gerardo, Monza, Lombardy, Italy